CLINICAL TRIAL: NCT00431821
Title: Reshaping Exercise Habits and Beliefs (REHAB): Pilot Testing of a Behavioral Intervention to Improve Mobility After Stroke
Brief Title: Reshaping Exercise Habits and Beliefs (REHAB)
Acronym: REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H24242
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Cerebrovascular Accident; Stroke
Keywords: Exercise; Rehabilitation; Stroke
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): Home-based exercise prescriptions with weekly motivational telephone calls.
  Interventions: Behavioral: Exercise
- Arm 2 (Other): Stroke education program with matched attention phone calls
  Interventions: Other: Stroke education

INTERVENTIONS:
Behavioral: Exercise — Home-based exercise prescriptions with weekly motivational telephone calls.
  Arms: Arm 1
Other: Stroke education — Stroke education program with matched attention phone calls
  Arms: Arm 2

SUMMARY:
Regular exercise has been demonstrated to improve muscle strength, balance, coordination as well as improve cardiovascular fitness levels and overall quality of life in stroke survivors. This study is designed to test the feasibility and effectiveness of a 12-week intervention to education and encourage stroke survivors to exercise following discharge from rehabilitation settings using a walking program and targeted functional activity homework.

ELIGIBILITY:
Inclusion Criteria:

1. 40-85 years old ischemic Stroke patients,
2. Stroke onset <90 days at enrollment,
3. Hemiparetic gait disorder,
4. Patients able to walk 30ft with or w/out assistive device,
5. Sufficient English comprehension to understand instructions, provide consent, and answer questions,
6. Lives within 30 miles of the Greater Baltimore area.

Exclusion Criteria:

1. Dementia (extended MMSE <85 or <80 if education level below 9th grade),
2. Untreated major clinical depression (CES-D>16) and confirmed with clinical interview,
3. Heavy alcohol use (<3 oz liquor, 3, 4-oz glasses of wine, or 3, 12- oz beers daily),
4. Active cancer, or any illness with a life expectancy of less than 6 months,
5. Any condition in which exercise activity would be contraindicated including, but not limited to: unstable angina, cardiac ischemic event within the past 6 months, congestive heart failure (Stage III or IV), major orthopedic chronic pain or non-stroke neuromuscular disorders restricting exercise, oxygen-dependent COPD or peripheral neuropathy.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-02 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Ambulatory Activity Profile | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Shaughnessy, RN PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251